CLINICAL TRIAL: NCT01686529
Title: Conjunctival Autografting Alone or Combined With Subconjunctival Bevacizumab for Primary Pterygium Treatment.
Brief Title: Bevacizumab for Primary Pterygium Treatment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Instituto de Oftalmología Fundación Conde de Valenciana (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: CC-008-2010
Record Dates: First submitted 2012-09-11; First posted 2012-09-18 (Estimated); Last update posted 2013-12-06 (Estimated); Status verified 2013-12

CONDITIONS: Pterygium
Keywords: Pterygium; bevacizumab; autoconjunctival graft
MeSH Terms: conditions — Pterygium | interventions — Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- One subconjunctival injection (Experimental): Autoconjunctival grafting and one subconjuntival bevacizumab injection (2.5mg/0.1ml) was applied after surgery
  Interventions: Procedure: Autoconjunctival grafting; Drug: Subconjuntival bevacizumab injection
- Two subconjuctival injections (Experimental): Autoconjunctival grafting and subconjuntival bevacizumab injection (2.5mg/0.1ml) was applied after surgery, with another injection 15 days after surgery
  Interventions: Procedure: Autoconjunctival grafting; Drug: Subconjuntival bevacizumab injection
- Conventional treatment (Active Comparator): Autoconjunctival grafting without subconjuntival bevacizumab injection
  Interventions: Procedure: Autoconjunctival grafting

INTERVENTIONS:
Procedure: Autoconjunctival grafting — The pterygium head was lifted off the corneal surface by blunt dissection. The pterygium body was dissected from the underlying sclera and thereafter excised. A thorough removal of Tenon's capsule was performed in an area much greater than the pterygium body. Free conjunctival autografting after pteryigum excision was performed as follows: the desired size of the conjunctiva under the upper eyelid was marked and excised. No limbal tissue was included in the graft. The excised tissue was placed on the bare sclera and tightly sutured to the sclera and the limbal area. Finally the autograft edges were sutured to the conjunctiva all around.
Drug: Subconjuntival bevacizumab injection — The subconjunctival injection of bevacizumab was applied adjacent to the site of pterygium separation inside the healthy conjunctiva. The half of the dose (1.25 mg/0.05ml) was applied in the nasal inferior quadrant, and the other half of the dose was applied in the nasal superior quadrant.
  Other Names: Avastin
  Arms: One subconjunctival injection; Two subconjuctival injections

SUMMARY:
The aim of this study was to investigate the efficacy and safety of subconjunctival bevacizumab application as an adjuvant therapy for primary pterygium.

ELIGIBILITY:
Inclusion Criteria:

* Patients with primary pterygium

Exclusion Criteria:

* Patients with diabetes mellitus
* collagenopathies,
* previous ocular surgeries,
* pregnant or lactating patients

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2010-03; Primary Completion 2011-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Pterygium recurrence | One point.
  The pterygium recurrence is evaluated at one year postoperative

SECONDARY OUTCOMES:
Conjunctival ischemia | Ischemia is measured at 24 h, 1 week, 15 days, six months and one year postoperative
  Whiteness of conjunctival bed, that means absence of blood vessels

CONTACTS AND LOCATIONS:
Overall Officials: Yonathan Garfias, MD, PhD, Principal Investigator — Instituto de Oftalmología
Locations (1):
- Instituto de Oftalmología, Mexico City, Mexico City, Mexico

REFERENCES:
- [Result] Nava-Castaneda A, Olvera-Morales O, Ramos-Castellon C, Garnica-Hayashi L, Garfias Y. Randomized, controlled trial of conjunctival autografting combined with subconjunctival bevacizumab for primary pterygium treatment: 1-year follow-up. Clin Exp Ophthalmol. 2014 Apr;42(3):235-41. doi: 10.1111/ceo.12140. Epub 2013 Jul 5. PMID 23777441
- See also: This is the link to the reference published on Pubmed — http://www.ncbi.nlm.nih.gov/pubmed/23777441